CLINICAL TRIAL: NCT02455713
Title: Effect of Positive Pressure Ventilation on Hemodynamics Around Delayed Sternal Closure Following Stage 1 Palliation of the Single Ventricle
Brief Title: Positive Pressure Ventilation and Sternal Closure in HLHS
Status: Withdrawn | Type: Observational
Why Stopped: Needed equipment failed before the study was started.
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Steven Schwartz, Professor of Paediatrics, The Hospital for Sick Children
Other Study IDs: 1000047473
Record Dates: First submitted 2015-04-05; First posted 2015-05-28 (Estimated); Last update posted 2018-05-01 (Actual); Status verified 2018-04

CONDITIONS: Hypoplastic Left Heart Syndrome
MeSH Terms: conditions — Hypoplastic Left Heart Syndrome | interventions — Positive-Pressure Respiration

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Intervention: Alter PEEP and PIP and measure hemodynamic outcomes.
  Interventions: Device: PEEP and PIP

INTERVENTIONS:
Device: PEEP and PIP — Changing ventilator settings and measuring oxygen delivery and cardiac output

SUMMARY:
This study will examine the cardiopulmonary interactions that occur with increasing ventilator settings (PEEP and PIP) in neonates after stage I palliation for hypoplastic left heart syndrome before and after sternal closure. Outcome measures include oxygen delivery and cardiac output.

DETAILED DESCRIPTION:
The objective of this study is to define the impact of variable levels of PEEP and tidal volume on hemodynamics and lung mechanics around delayed sternal closure after Stage 1 palliation in the single ventricle patient.

The Specific Aims of this work are:

Specific Aim 1: Evaluate hemodynamics and lung mechanics across a range of PEEP (2-12 cm H2O) before and after chest closure, while maintaining consistent ventilation, in infants with single ventricle physiology who undergo delayed sternal closure after Stage 1 palliation surgery.

Specific Aim 2: Evaluate hemodynamics and lung mechanics across a range of tidal volumes (6-15ml/kg) and before and after chest closure, while maintaining consistent ventilation, in infants with single ventricle physiology who undergo delayed sternal closure after Stage 1 palliation surgery.

Hypotheses

1. The effects of PEEP and tidal volume on hemodynamics and lung mechanics will be significantly different before and after sternal closure. We expect that there will be little effect of PEEP or tidal volume when the sternum remains open. Once the sternum is closed, we hypothesize that those with shunted single ventricle physiology will have optimal oxygen delivery and lung mechanics with modest PEEP and tidal volume (U-shaped curves).

Rationale: Delayed sternal closure is commonly used to prevent tissue tamponade and promote favorable hemodynamics in critically ill patients following surgery for congenital heart disease. This technique is frequently employed in shunted single ventricle physiology (i.e.- Norwood patients). While there have been several studies that have shown that sternal closure is associated with temporary hemodynamic changes and stiffer lung mechanics, there have been no prospective studies of the impact of different ventilator strategies on hemodynamics, and lung mechanics before and after sternal closure. Because these patients are generally among the most fragile postoperative patients, it is critical to understand if specific ventilator strategies can help mitigate any negative hemodynamic consequences of chest closure. The purpose of this study is to understand the critical cardiopulmonary interactions that occur with delayed sternal closure in this population, and to determine optimal approaches to mechanical ventilation under these different circumstances.

Cardiopulmonary interactions differ based on the underlying cardiac anatomy and physiology. Most studies of cardiopulmonary interactions following surgery for congenital heart disease have examined the difference between positive and negative pressure ventilation in those with right ventricular restrictive physiology such as after tetralogy of Fallot repair, or after cavopulmonary connection surgery. This work consistently shows improvement in cardiac output and pulmonary blood flow with negative pressure ventilation. It is not practical, however, to maintain negative pressure ventilation when the sternum remains open and it is not even clear that the same cardiopulmonary interactions are at play in the absence of significant elastic recoil forces of the chest wall.

Similarly, while patients with left ventricular dysfunction generally benefit from positive pressure ventilation, there is no data regarding the hemodynamic effects of positive pressure ventilation in left ventricular dysfunction when intrathoracic pressure will not deviate from atmospheric, which is the situation with delayed sternal closure.

Shunted single ventricle physiology is perhaps the most difficult for which to predict the effects of different ventilator strategies before and after sternal closure. The combination of parallel pulmonary and systemic circulations, less than optimal total cardiac output and, most commonly, at least some pulmonary edema make it difficult to predict the ideal ventilator strategy. Studies in this population have focused more on the effects of FiO2 and hyperventilation than on respiratory mechanics and cardiopulmonary interactions. Nevertheless, this work has shown that the occurrence of pulmonary venous desaturation is common following stage 1 Norwood surgery, and it remains unknown if there is risk or benefit from strategies such as lower or higher tidal volumes or lower or higher PEEP on hemodynamics and oxygen delivery.

ELIGIBILITY:
Inclusion Criteria:

1. All patients who, following stage 1 palliation for single ventricle physiology, undergo delayed sternal closure are eligible to be included in the study

Exclusion Criteria:

1. History of pneumothorax, acute respiratory distress syndrome, or other contraindication to the proposed ventilator manipulations as determined by the responsible CCCU staff physician.
2. Endotracheal tube leak > 15%.
3. Lack of informed consent from parents.
4. Weight less than 2.6kg

Max Age: 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants after congenital heart surgery.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2015-02; Primary Completion 2016-12 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Oxygen Delivery calculated from direct measurements of oxygen consumption via respiratory mass spectrometry | Measurements made 15 minutes after each ventilator change. Total duration of observation is 2.5 hours.
  Oxygen delivery will be calculated from direct measurements of oxygen consumption via respiratory mass spectrometry and estimates of cardiac output calculated using the Fick equation from measured arterial a venous blood gas samples.

SECONDARY OUTCOMES:
Cardiac Output calculated using the Fick Equation | Measurements made 15 minutes after each ventilator change. Total duration of observation is 2.5 hours.
  Cardiac output will be calculated using the Fick Equation from direct measurement of oxygen consumption using respiratory mass spectrometry and arterial and venous blood gas samples.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Schwartz, MD, Principal Investigator — The Hospital for Sick Children, Toronto
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada